CLINICAL TRIAL: NCT03891992
Title: Role of High Resolution Ultrasound Imaging in Evaluation of Shoulder Pain Guided by Magnetic Resonance Imaging Findings
Brief Title: High Resolution Ultrasound in Evaluation of Shoulder Pain Guided by MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shehab Gamal Abdallah, principal investigator, Assiut University
Other Study IDs: ultrasound in shoulder pain
Record Dates: First submitted 2019-03-15; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To asses causes of shoulder pain by Ultrasound in guide of MRI diagnosis to help Ultrasound to be used alone in the future

DETAILED DESCRIPTION:
shoulder pain is a common medical condition, particularly in middle-aged and older adults, Shoulder pain makes up about 15% of all musculoskeletal complaints and has an incidence of 25 cases/1000 patients from 45-64 years old. Most shoulder problems fall into three major categories: soft tissue disorders, articular injury or instability, and arthritis. The incidence of lesions increases with age as tendon tissue progressively weakens or degenerates, but repeated microtrauma or overuse from professional or athletic activity can also cause soft tissue problems in all age groups.Patients younger than 30 yrs. old tend to have mild inflammatory or biomechanical causes for their pain such as a traumatic instability, tendinosis and arthropathy.The major cause of shoulder pain in patients older than 40 years is rotator cuff impingement and tears.There are no clear national guidelines for the diagnosis of shoulder pain. Several diagnostic tests are used for the diagnosis of soft tissue disorders, including clinical assessment, ultrasonography, magnetic resonance imaging (MRI), CT , X-ray and Arthroscopy. Shoulder pain is common, but the complexity of the shoulder joint frequently creates a diagnostic challenge for clinicians trying to identify the source of pain. As it is the most mobile joint in the body, the shoulder has a wide variety of physical exam maneuvers and tests designed to help the clinician diagnose shoulder pathology. So the current challenge from the clinicians is to understand which physical exam test(s) can provide sensitive and specific data to diagnose shoulder pathology. Evaluation of these exam maneuvers is of moderate to low quality, but still provides valuable information on how to interpret these exam results. Ultrasound , In addition to the physical exam, point-of care diagnostic musculoskeletal ultrasound has evolved as a useful and powerful tool for both diagnosis and treatment of shoulder pain, and it has many advantages like being relatively inexpensive, noninvasive and widely available.Ultrasound is increasingly being used to image many of the structures that can cause chronic shoulder pain. Ultrasound has excellent in-plane and beam-thickness spatial resolution , although the contrast resolution of many abnormalities in the shoulder is less than that with MRI, and also it is particularly useful in patients with a suspected supraspinatus or infraspinatus tendon tear, but is also helpful in the assessment of the subscapularis, acromioclavicular joint capsule and osteophytes, biceps tendon, subacromial-subdeltoid bursa, and the spinoglenoid notch. Ultrasound also allows dynamic imaging, which can be helpful when looking for biceps tendon subluxation, subscapularis tendon tears, and arm-abduction supraspinatus tendon impingement .

ELIGIBILITY:
Inclusion Criteria:

* Patients. have positive tests of shoulder pain by clinical examination.
* Patients who suspected by Plain X-ray to have shoulder instability.

Exclusion Criteria:

* Patients who previously underwent surgical intervention to shoulder joint for any reason.
* Patients with history of fracture repaired by metal plates or screws.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients have positive tests of shoulder pain by clinical examination and suspected by Plain X-ray to have shoulder instability.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
ultrasound findings in shoulder pain | baseline
  to see if the same findings found by magnetic resonance in cases of shoulder pain imaging will appear by high resolution ultrasound

IPD SHARING:
Plan to Share IPD: Undecided